CLINICAL TRIAL: NCT02584101
Title: The Use of Acceptance and Commitment Therapy to Promote WellBeing and Psychological Flexibility in Carers: A Randomized Controlled Feasibility Trial
Brief Title: Acceptance and Commitment Therapy (ACT) and Carers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Glasgow (Other)
Collaborators: Brain Injury Rehabilitation Trust (Other)
Responsible Party: Principal Investigator, Ross White, Senior Lecturer, University of Glasgow
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 15/WS/0208
Record Dates: First submitted 2015-10-21; First posted 2015-10-22 (Estimated); Last update posted 2016-05-26 (Estimated); Status verified 2016-05

CONDITIONS: Brain Injuries
Keywords: Acceptance and Commitment Therapy
MeSH Terms: conditions — Brain Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- ACT (Experimental): ACT therapy
  Interventions: Behavioral: ACT
- Enhanced Treatment as Usual (Active Comparator): Group support
  Interventions: Behavioral: Enhanced Treatment as Usual

INTERVENTIONS:
Behavioral: ACT — ACT therapy administered in 3 sessions over a 4 week period
  Arms: ACT
Behavioral: Enhanced Treatment as Usual — 2 group discussion sessions over a 4 week period
  Arms: Enhanced Treatment as Usual

SUMMARY:
Background: Research has extensively documented the adverse impact that caring for an individual with an acquired brain injury can have including financial difficulties, social isolation, family tension and conflict, relationship difficulties, role adjustment and psychological distress (Foster et al., 2012). Research has indicated that Acceptance and Commitment Therapy (ACT) shows promise for increasing wellbeing and psychological flexibility in caregivers and could be a useful intervention for use with this population.

Aims: The primary aim of this study is to investigate the feasibility of using an ACT intervention to enhance the wellbeing and the psychological flexibility of carers using the Population, Intervention, Control, and Outcomes (PICO) framework. Methods: The current study is a randomised control design, exploring the feasibility of comparing the efficacy of an ACT intervention to Enhanced Treatment As Usual (ETAU), to improve the wellbeing of the carers of adults with an acquired brain injury (ABI). Participants will be recruited from the Brain Injury Rehabilitation Trust (BIRT) in Glasgow, Scotland and randomly assigned to either an ACT intervention group or TAU control group. Both will be assessed in parallel to one another completing a range of baseline and post-baseline measures. Applications: This feasibility study will provide information for further research on the utilisation of an ACT intervention to improve the wellbeing of carers and whether this is an acceptable intervention for this population.

ELIGIBILITY:
Inclusion Criteria:

* full time or part time carer for an adult with an acquired brain injury

Exclusion Criteria:

* learning disability
* not proficient in English

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2016-01; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Well-being | 4 weeks
  Change in General Health Questionnaire (GHQ-12) score

SECONDARY OUTCOMES:
Psychological Flexibility | 4 weeks
  Change in Acceptance and Action Questionnaire (AAQII) score
Values | 4 weeks
  Change in Valuing Questionnaire (VQ) score
Experiential Avoidance | 4 weeks
  Change in Experiential Avoidance in Caregiving Questionnaire (EACQ) score

CONTACTS AND LOCATIONS:
Overall Officials: Ross White, BSc(Hons) PhD DClinPsy, Principal Investigator — University of Glasgow
Locations (1):
- Brain Injury Rehabilitation Trust, Glasgow, United Kingdom